CLINICAL TRIAL: NCT03037151
Title: Safety and Fibrosis Improvement of Grazoprevir and Elbasvir for HCV GT1 and GT6 With or Without HIV
Brief Title: Safety and Efficacy of Grazoprevir and Elbasvir for GT1ang GT6 With and Without HIV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Chulalongkorn University (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIV-NAT 245
Record Dates: First submitted 2017-01-27; First posted 2017-01-31 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Compensated Cirrhosis
Keywords: Safety; Efficacy; grazoprevir; elbasvir; compensated cirrhosis; genotype 1 (GT1); genotype 6 (GT6); hepatitis virus C (HCV); human immunodeficiency virus (HIV)
MeSH Terms: conditions — Hepatitis C; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HCV mono-infection Treatment naives (Experimental): HCV treatment-naïve patients will be treated with the combination of grazoprevir plus elbasvir for 12 weeks.
  Interventions: Drug: Grazaoprevir/Elbasavir
- HCV mono-infection Treatment experienced (Experimental): HCV treatment-experienced patients, including null responders, partial responders or post-treatment relapsers, will be assigned to treat with the combination plus weight-based RBV for 16 weeks.
  Interventions: Drug: Grazaoprevir/Elbasavir/RBV
- HCV/HIV co-infection Treatment naives (Experimental): HCV/HIV coinfected, treatment-naïve patients will be treated with the combination of grazoprevir plus elbasvir for 12 weeks.
  Interventions: Drug: Grazaoprevir/Elbasavir
- HCV/HIV co-infection Treatment experienced (Experimental): HCV/HIV co-infected treatment-experienced patients, including null responders, partial responders or post-treatment relapsers, will be assigned to treat with the combination plus weight-based RBV for 16 weeks.
  Interventions: Drug: Grazaoprevir/Elbasavir/RBV

INTERVENTIONS:
Drug: Grazaoprevir/Elbasavir — treatment naive
  Arms: HCV mono-infection Treatment naives; HCV/HIV co-infection Treatment naives
Drug: Grazaoprevir/Elbasavir/RBV — treatment experienced
  Arms: HCV mono-infection Treatment experienced; HCV/HIV co-infection Treatment experienced

SUMMARY:
This study will evaluate the safety and efficacy of combination treatment with grazoprevir + elbasvir for compensated cirrhotic participants with chronic genotype 1 (GT1) and genotype 6 (GT6) hepatitis C virus (HCV) infection with or without human immunodeficiency virus (HIV) infection.

DETAILED DESCRIPTION:
Total 100 patients with compensated cirrhosis, chronically infected with HCV GT1 or GT6 with or without HIV infection will be included. Patients with HCV GT1 and GT6 will be enrolled on a 1:1 basis (approximately 50 patients with GT1 and 50 patients with GT6). Treatment-naïve patients will be treated with the combination of grazoprevir plus elbasvir for 12 weeks. Treatment-experienced patients, including null responders, partial responders or post-treatment relapsers, will be assigned to treat with the combination plus weight-based RBV for 16 weeks. The dosages of study drugs are 100 mg of grazoprevir once daily and 50 mg of elbasvir once daily. All patients will follow up to assess SVR (defined by HCV RNA level <12 IU/mL) at week12 and week 24 after treatment (SVR12 and SVR24, respectively). Additionally, participants will be evaluated the longitudinal changes in LS values by TE up to 240 weeks (5 years) after treatment

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 years or older
2. Documented chronic HCV GT1 or GT6 (positive for anti-HCV antibody and HCV RNA at least 6 months prior to screening)
3. HCV RNA of at least 10,000 IU/ml
4. Cirrhosis defined by: liver biopsy showing cirrhosis METAVIR F4; or TE showing cirrhosis with a result of >13.0 kPa
5. Treatment-naïve individuals for chronic HCV infection
6. Treatment-experienced individuals (Previous treatment failure with PEG-IFN plus RBV) for chronic HCV infection
7. HIV-infected participants enrolled in this study must meet following criteria:

   7.1 Documented HIV infection 7.2 Naïve to treatment with any antiretroviral therapy (ART) or on HIV ART for at least 8 weeks prior to study entry using a dual nucleoside reverse transcriptase inhibitor (NRTI) backbone of tenofovir or abacavir and either emtricitabine or lamivudine plus raltegravir (or dolutegravir or rilpivirine) 7.3 CD4+ T-cell count >200 cells/mm3 if on ART or >500 cell/mm3 if ART treatment naïve 7.4 Undetectable plasma HIV-RNA at least 8 weeks prior to screening if on ART or <50,000 copies/mL if ART treatment naïve
8. Agree to use two acceptable methods of birth control from at least 2 weeks prior to Day 1 and continue until at least 6 months after last dose of study drug, or longer if dictated by local regulations (for female subject who is of childbearing potential or male subject with female sexual partner who is of childbearing potential).

Exclusion Criteria:

1. Evidence of decompensated liver disease (Child-Pugh Class B or C or Child-Pugh score >6, platelets less than 75 × 10³/μL, serum albumin < 3·0 g/dL, presence of or history of ascites, gastric or variceal bleeding, hepatic encephalopathy or other signs or symptoms of advanced liver disease)
2. Co-infected with hepatitis B virus
3. Has cirrhosis and liver imaging within 6 months showing evidence of HCC or is under evaluation for HCC
4. Pregnant or breast-feeding from day 1 or anytime during treatment, and 14 days after the last dose of study medication
5. Any medical condition requiring or likely to require chronic systemic administration of corticosteroids or other immunosuppressant drugs during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of SVR12 | 12 weeks post-treatment
  To evaluate the rate of sustained virological response (SVR) at 12 weeks after the end of treatment (SVR12) in compensated cirrhotic participants with GT1 and GT6 HCV infection with or without HIV infection treated with the combination of grazoprevir and elbasvir

SECONDARY OUTCOMES:
Rate of SVR24 | 24 weeks post-treatment
  To evaluate the rate of sustained virological response (SVR) at 24 weeks after the end of treatment (SVR24)
Decline of liver stiffness | 5 years post-treatment
  To evaluate the percentage of participants achieving a significant decline in liver stiffness (LS) values (defined as a ≥30% decrease from baseline) up to 240 weeks (5 years) after treatment
changes in liver stiffness | 5 years
  To compare the longitudinal changes in LS values over time between participants and untreated historical controls

CONTACTS AND LOCATIONS:
Overall Officials: Anchalee Avihingsanon, MD, PhD, Principal Investigator — HIV-NAT, Thai Red Cross - AIDS Research Centre; Pisit Tangkijvanich, MD, Principal Investigator — Chulalongkorn University
Locations (2):
- Thailand (2):
  - Faculty of Medicine, Chulalongkorn University, Bangkok
  - HIV-NAT, Thai Red Cross AIDS Research Centre, Bangkok

IPD SHARING:
Plan to Share IPD: No
only when needed as per the auditing/monitoring processes and requirement

REFERENCES:
- See also: Related Info — http://www.hivnat.org